CLINICAL TRIAL: NCT01587651
Title: A Pharmacodynamic Evaluation of Switching From Ticagrelor to Prasugrel in Subjects With Stable Coronary Artery Disease: 2nd Switching Antiplatelet Agents
Brief Title: Pharmacodynamic Evaluation of Switching From Ticagrelor to Prasugrel in Subjects With Stable Coronary Artery Disease
Acronym: SWAP-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS747s-B-U4003
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: CAD; prasugrel; ticagrelor; antiplatelet; thienopyridine; P2Y12 Inhibitors
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prasugrel Maintenance Dose (Experimental): Prasugrel 10 mg QD MD
  Interventions: Drug: Prasugrel Maintenance Dose
- Ticagrelor Maintenance Dose (Active Comparator): Ticagrelor 90 mg twice-daily (BID) MD
  Interventions: Drug: Ticagrelor Maintenance Dose
- Prasugrel Loading Dose (Experimental): Prasugrel 60mg Loading Dose (LD), followed by prasugrel 10mg once-daily (QD) Maintenance Dose (MD)
  Interventions: Drug: Prasugrel Loading Dose; Drug: Prasugrel Maintenance Dose

INTERVENTIONS:
Drug: Prasugrel Loading Dose — 60mg given as six 10mg film coated tablets
  Other Names: Effient
  Arms: Prasugrel Loading Dose
Drug: Prasugrel Maintenance Dose — 10mg maintenance dose, given as one 10mg film coated tablet
  Other Names: Effient
  Arms: Prasugrel Loading Dose; Prasugrel Maintenance Dose
Drug: Ticagrelor Maintenance Dose — one 90mg film coated tablet
  Other Names: Brilinta
  Arms: Ticagrelor Maintenance Dose

SUMMARY:
This is a Phase 4, multicenter, open-label (blinded Pharmacodynamic PD results), randomized, 3-arm, parallel-design study of subjects with stable Coronary Artery Disease CAD. This study will compare the PD effect of prasugrel 10 mg QD (once-daily) maintenance dose with ticagrelor 90 mg BID (twice daily) maintenance dose in subjects with stable CAD who have previously received ticagrelor loading does (LD) and maintenance dose (MD)..

ELIGIBILITY:
Inclusion Criteria:

* Male or female; age >= 18 and < 75 years
* Weight >= 60 kg
* Receiving low dose ASA (75 mg to 150 mg daily) for at least 7 days at the time of Visit 1 and able to continue the same regimen throughout the study
* Stable CAD. CAD is defined as any of the following:
* History of a positive stress test
* Previous coronary revascularization including percutaneous coronary intervention (PCI), stent, or coronary artery bypass graft (CABG)
* Angiographic demonstration of CAD (at least

  1 lesion >= 50 percent)
* Presence of at least moderate plaque by computed tomography (CT) angiography
* Electron beam CT coronary artery calcification score >= 100 Agatston units
* If female, may be enrolled if

One of the following 3 criteria are met:

* Had a hysterectomy or tubal ligation at least 6 months prior to signing the informed consent form (ICF)
* Post-menopausal for at least 1 year
* If of childbearing potential, will practice 1 of the following methods of birth control throughout the study: oral, injectable, or implantable hormonal contraceptives; intrauterine device; diaphragm plus spermicide; or female condom plus spermicide. Methods of contraception that are not acceptable are partner's use of condoms or partner's vasectomy
* Able and willing to provide written informed consent before entering the study

Exclusion Criteria:

* Have a defined need for adenosine diphosphate (ADP)-receptor inhibitor therapy, such as any of the following (or any other condition that in the Investigator's judgment would require such therapy):
* Within =< 12 months of an acute coronary syndrome (ACS) event (unstable angina [UA], non-ST-elevation myocardial infarction [NSTEMI], or ST-elevation myocardial infarction [STEMI]) regardless of initial treatment (that is, invasive versus noninvasive)
* Subjects who underwent angioplasty within 12 months including bare-metal stent and/or a drug-eluting stent
* Had any stent placed in an unprotected left main coronary artery or in the last patent artery within the last 12 months
* Received thienopyridine therapy within 30 days of study entry
* Plan to undergo coronary revascularization at any time during the trial
* Presence or history of any of the following: ischemic or hemorrhagic stroke; transient ischemic attack (TIA); intracranial neoplasm; arteriovenous malformation, or aneurysm; intracranial hemorrhage; head trauma (within 3 months of study entry)
* History of refractory ventricular arrhythmias with an increased risk of bradycardic events (eg, subjects without a pacemaker who have sick sinus syndrome, 2nd or 3rd degree atrioventricular (AV) block or bradycardic-related syncope)
* History or evidence of congestive heart failure (New York Heart Association Class III or above =< 6 months before screening
* Severe hepatic impairment
* History of uric acid nephropathy
* Uncontrolled hypertension, or systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg at screening
* Severely impaired renal function (glomerular filtration rate < 30 mL/minute) or on dialysis
* At risk for bleeding
* Taking prohibited medications

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (8):
  - Univ. of Florida College Medicine, Jacksonville, Florida
  - Clinical Pharmacology Unit of Miami, Miami, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Sinai Center for Thrombosis Research, Baltimore, Maryland
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - West Houston Area Clinical Trial Consultants, Houston, Texas
  - Cardiology Center of Houston, Katy, Texas
- United Kingdom (5):
  - University Hospital of Wales, Heathpark, Cardiff
  - Bristol Heart Institute, Bristol
  - University Hospital Leicester, Leicester
  - Southampton General Hospital, Southampton
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects must have been taking low dose aspirin (ASA) (75 mg to 150 mg once daily-QD) for at least 7 days prior to Screening (Visit 1), and must have continued the same regimen throughout the study.
Pre-assignment Details: The study consisted of a 3 to 5 day ticagrelor run-in phase followed by randomized treatment on 1 of 2 prasugrel regimens or continued ticagrelor
Groups:
- Prasugrel Loading Dose: Prasugrel 60mg Loading Dose (LD), followed by prasugrel 10mg once-daily (QD) Maintenance Dose (MD)
  Prasugrel Maintenance Dose : 10mg maintenance dose, given as one 10mg film coated tablet
  Prasugrel Loading Dose : 60mg given as six 10mg film coated tablets
- Prasugrel Maintenance Dose: Prasugrel 10 mg QD MD
  Prasugrel Maintenance Dose : 10mg maintenance dose, given as one 10mg film coated tablet
- Ticagrelor Maintenance Dose: Ticagrelor 90 mg twice-daily (BID) MD
  Ticagrelor Maintenance Dose : one 90mg film coated tablet
Period: Overall Study
Arm/Group | Prasugrel Loading Dose | Prasugrel Maintenance Dose | Ticagrelor Maintenance Dose
Started | 34 | 41 | 35
Completed | 34 | 38 | 34
Not Completed | 0 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel Loading Dose | Prasugrel Maintenance Dose | Ticagrelor Maintenance Dose | Total
Number analyzed (Participants) | 34 | 41 | 35 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 28 | 22 | 74
  >=65 years | 10 | 13 | 13 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.69) | 58.5 (8.84) | 61.5 (6.87) | 59.2 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 8 | 29
  Male | 24 | 30 | 27 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4 | 8
  Not Hispanic or Latino | 33 | 36 | 30 | 99
  Unknown or Not Reported | 0 | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 4 | 18
  White | 26 | 33 | 30 | 89
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 36 | 32 | 98
  United Kingdom | 4 | 5 | 3 | 12
weight [Mean (Standard Deviation); unit: kg] | 97.0 (17.70) | 95.4 (18.85) | 89.4 (19.35) | 94.0 (18.77)
height [Mean (Standard Deviation); unit: cm] | 171.2 (8.74) | 171.9 (10.15) | 174.3 (9.14) | 172.4 (9.41)
body mass index [Mean (Standard Deviation); unit: kg/m^2] | 33.2 (5.88) | 32.3 (5.92) | 29.2 (4.82) | 31.6 (5.77)
diabetes mellitus history [Number; unit: participants] — number of participants with diabetes mellitus sum of categories does not equal number of participants due to not all participants having this specific medical condition
  participants | 14 | 12 | 5 | 31
hypertension history [Number; unit: participants] — number of participants with hypertension susum of categories does not equal number of participants due to not all participants having this specific medical condition
  participants | 26 | 29 | 24 | 79
hyperlipidemia history [Number; unit: participants] — number of participants with hyperlipidemia sum of categories does not equal number of participants due to not all participants having this specific medical condition
  participants | 32 | 35 | 31 | 98
peripheral artery disease history [Number; unit: participants] — number of participants with peripheral artery disease (PAD) sum of categories does not equal number of participants due to not all participants having this specific medical condition
  participants | 2 | 1 | 2 | 5
body mass index category [Number; unit: participants] — body mass index <30 kg/m^2 or >= 30 kg/m^2 sum of categories does not equal number of participants due to missing data for 1 subject
  participants
    < 30 kg/m^2 | 13 | 16 | 24 | 53
    >= 30 kg/m^2 | 21 | 24 | 11 | 56
    Unknown | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Units
Description: P2Y12 Reaction Units (PRU) measured by VerifyNow P2Y12 assay VerifyNow P2Y12 assay, developed by Accumetrics, Inc. (San Diego, CA, USA), has been approved by the FDA to assess clopidogrel response using whole blood in a point-of-care testing fashion. Platelet aggregation with this system is defined by PRU, with a higher PRU indicative of greater platelet aggregation, and a lower PRU indicative of inhibition.
Time Frame: 7 days after first randomized dose
Population: Primary Population includes all subjects who received at least 1 dose of randomized study drug and have valid PRU data at both randomization visit pre-dosing and end-of-treatment visit. A subject is considered to have valid PRU data for primary PD analyses if he/she does not have certain protocol deviations listed in Statistical Analysis Plan.
Measure: Least Squares Mean (Standard Error); unit: PRU (P2Y12 Reaction Units)
Groups:
- Prasugrel Combined Groups: combined Prasugrel loading dose and Prasugrel maintenance dose
Arm/Group | Prasugrel Combined Groups | Ticagrelor
Number analyzed (Participants) | 65 | 33
PRU (P2Y12 Reaction Units) | 95.0 (6.18) | 49.0 (8.68)
Statistical Analysis 1: Comparison: Prasugrel Combined Groups vs Ticagrelor; ANCOVA model included treatment as a main effect and pre-randomization baseline PRU as a covariate. The combined prasugrel groups were modeled as a single treatment. If the upper limit of the CI for the mean difference was not greater than 45 PRU, then the PD response to prasugrel 10 mg QD MD was deemed noninferior to that achieved by ticagrelor 90 mg BID MD; Test type: Non-Inferiority or Equivalence — Noninferiority was assessed using a 95% CI of the difference in mean PRU between ticagrelor and prasugrel (2 arms combined). Under the assumption of 0 difference in mean PRU between prasugrel 10 mg QD MD and ticagrelor 90 mg BID MD, a common SD of 60 PRU (based on previous DSI studies and published data), and a drop-out rate not exceeding 15%, a sample size of 105 allows for the 95% CI to stay within ± 45 PRU (non-inferiority margin) with a power of 90%; Mean Difference (Final Values) = 46.0, 95% CI 2-sided [24.9 to 67.2], Standard Error of Mean 10.66

2. Secondary Outcome: P2Y12 Reaction Units
Description: P2Y12 Reaction Units (PRU) measured by VerifyNow P2Y12 assay measured at 2, 4, 24, 48 hours after first randomized study treatment
Time Frame: 2, 4, 24, 48 hours after first randomized dose
Population: Primary Population
Measure: Least Squares Mean (Standard Error); unit: PRU
Groups:
- Prasugrel Loading Dose: prasugrel 60 mg loading dose followed by 10 mg QD for 6 days
- Prasugrel Maintenance Dose: prasugrel 10 mg QD for 7 days
Arm/Group | Prasugrel Combined Groups | Ticagrelor | Prasugrel Loading Dose | Prasugrel Maintenance Dose
Number analyzed (Participants) | 65 | 33 | 31 | 34
PRU
  2 hours | 33.7 (3.18) | 28.9 (4.24) | 22.1 (4.22) | 44.8 (4.15)
  4 hours | 41.1 (3.67) | 29.3 (4.54) | 24.1 (4.69) | 57.0 (4.53)
  24 hours | 126.8 (7.57) | 47.6 (8.71) | 81.6 (8.86) | 167.8 (8.44)
  48 hours | 159.3 (7.68) | 38.6 (9.07) | 118.3 (9.22) | 199.0 (9.07)

3. Secondary Outcome: Platelet Reactivity Index
Description: Platelet Reactivity Index (PRI) by the Vasodilator-Stimulated Phosphoprotein(VASP) assay 2, 4, 24, 48 hours and 7 days after first randomized study treatment.
  The VASP assay is an indirect, but relatively specific measure of inhibition of P2Y12-induced platelet activation. The assay quantifies the level of phosphorylation of the intracellular protein VASP, which undergoes phosphorylation when platelet P2Y12 receptors are blocked. The level of VASP phosphorylation, expressed as the PRI, represents the percentage inhibition relative to an assay baseline/maximal P2Y12-independent platelet aggregation.
Time Frame: 2, 4, 24, 48 hours, 7 days after first randomized dose
Population: Primary Population
Measure: Least Squares Mean (Standard Error); unit: percentage PRI
Arm/Group | Prasugrel Combined Groups | Ticagrelor | Prasugrel Loading Dose | Prasugrel Maintenance Dose
Number analyzed (Participants) | 65 | 33 | 31 | 34
percentage PRI
  2 hours post-dose | 18.2 (1.37) | 13.2 (1.85) | 15.8 (1.94) | 20.4 (1.87)
  4 hours post-dose | 16.3 (1.58) | 14.3 (2.06) | 11.4 (2.16) | 20.9 (2.08)
  24 hours post-dose | 34.3 (2.24) | 19.1 (2.71) | 24.2 (2.85) | 43.7 (2.74)
  48 hours post-dose | 48.1 (2.58) | 18.7 (3.20) | 38.0 (3.37) | 57.7 (3.30)
  7 days post-dose | 33.5 (2.64) | 19.8 (3.58) | 38.8 (3.87) | 29.1 (3.50)

4. Secondary Outcome: PRU Percent Inhibition (Device-reported)
Description: PRU VerifyNow P2Y12 assay device-reported percent inhibition 2, 4, 24, and 48 hours, and 7 days after first randomized study treatment
  VerifyNow P2Y12 assay, developed by Accumetrics, Inc. (San Diego, CA, USA), has been approved by the FDA to assess clopidogrel response using whole blood in a point-of-care testing fashion. The percent inhibition reported by VerifyNow device represents the percentage inhibition relative to maximal P2Y12-independent platelet aggregation achieved with the same sample in the presence of the iso-thrombin receptor activating peptide.
Time Frame: 2, 4, 24, 48 hours, 7 days after first randomized dose
Population: Primary population
Measure: Least Squares Mean (Standard Error); unit: percent inhibition
Arm/Group | Prasugrel Combined Groups | Ticagrelor | Prasugrel Loading Dose | Prasugrel Maintenance Dose
Number analyzed (Participants) | 65 | 33 | 31 | 34
percent inhibition
  2 hours post-dose | 87.8 (1.13) | 89.2 (1.53) | 91.4 (1.53) | 84.3 (1.51)
  4 hours post-dose | 84.9 (1.25) | 89.6 (1.58) | 90.2 (1.63) | 79.8 (1.58)
  24 hours post-dose | 54.1 (2.68) | 81.9 (3.13) | 69.6 (3.18) | 40.0 (3.03)
  48 hours post-dose | 42.3 (2.79) | 85.8 (3.19) | 58.3 (3.24) | 26.8 (3.19)
  7 days post-dose | 65.5 (2.17) | 81.0 (3.07) | 65.6 (3.16) | 65.4 (3.02)

5. Secondary Outcome: PRU Percent Inhibition (Calculated)
Description: Analysis of Mean Calculated Percent Inhibition by time point
  Calculated percent inhibition at time point t is defined as: 100 × (baseline PRU - PRUt)/baseline PRU where baseline PRU is the VerifyNow PRU value at pre-run-in baseline and PRUt is the VerifyNow PRU value at time t.
Time Frame: 2, 4, 24, 48 hours, 7 days after first randomized dose
Population: Primary population
Measure: Least Squares Mean (Standard Error); unit: Percent Inhibition
Arm/Group | Prasugrel Combined Groups | Ticagrelor | Prasugrel Loading Dose | Prasugrel Maintenance Dose
Number analyzed (Participants) | 65 | 33 | 31 | 34
Percent Inhibition
  2 hours post-dose | 88.22 (1.113) | 89.73 (1.476) | 92.55 (1.475) | 84.15 (1.429)
  4 hours post dose | 85.06 (1.319) | 89.26 (1.632) | 91.36 (1.686) | 79.35 (1.605)
  24 hours post dose | 53.63 (2.851) | 81.86 (3.237) | 71.40 (3.291) | 38.01 (3.085)
  48 hours post dose | 41.59 (2.911) | 85.06 (3.388) | 57.98 (3.438) | 26.20 (3.332)
  7 days psot dose | 64.97 (2.336) | 80.69 (3.322) | 64.97 (3.429) | 64.97 (3.221)

6. Secondary Outcome: Percentage of Subjects With High On-treatment Platelet Reactivity
Description: Percentage of subjects with High on-treatment Platelet Reactivity (HPR) defined as a) >= 208 PRU and b) >= 230 PRU by the VerifyNow P2Y12 assay and c) >50% PRI by the VASP assay, 2, 4, 24, and 48 hours and 7 days after first randomized study treatment.
  A poor response of the platelets to "drug", called High Residual Platelet Reactivity (HRPR), has been incriminated to account for a recurrence of ischemic events
Time Frame: 2, 4, 24, 48 hours, 7 days after first randomized dose
Population: Primary population
Measure: Number; unit: percentage of subjects
Arm/Group | Prasugrel Combined Groups | Ticagrelor | Prasugrel Loading Dose | Prasugrel Maintenance Dose
Number analyzed (Participants) | 65 | 33 | 31 | 34
percentage of subjects
  >= 208 PRU 2 hours post dose | 0 | 0 | 0 | 0
  >= 208 PRU 4 hours post dose | 0 | 0 | 0 | 0
  >= 208 PRU 24 hours post dose | 17.5 | 0 | 3.3 | 37.5
  >= 208 PRU 48 hours post dose | 30.2 | 0 | 16.1 | 43.8
  >= 208 PRU 7 days post dose | 1.5 | 3 | 3.2 | 0
  >= 230 PRU by VerifyNow P2Y12 2 hours post dose | 0 | 0 | 0 | 0
  >= 230 PRU by VerifyNow P2Y12 4 hours post dose | 0 | 0 | 0 | 0
  >= 230 PRU by VerifyNow P2Y12 24 hours post dose | 14.3 | 0 | 3.3 | 24.2
  >= 230 PRU by VerifyNow P2Y12 48 hours post dose | 22.2 | 0 | 6.5 | 37.5
  >= 230 PRU by VerifyNow P2Y12 7 days post dose | 1.5 | 3 | 3.2 | 0
  >50% PRI by VASP assay 2 hours post dose | 3.5 | 3.3 | 3.6 | 3.4
  >50% PRI by VASP assay 4 hours post dose | 1.8 | 3.3 | 0 | 3.4
  >50% PRI by VASP assay 24 hours post dose | 21.3 | 12.9 | 3.4 | 37.5
  >50% PRI by VASP assay 48 hours post dose | 45 | 6.3 | 13.8 | 74.2
  >50% PRI by VASP assay 7 days post dose | 15.5 | 3.4 | 23.1 | 9.4

ADVERSE EVENTS:
Arm/Group | Prasugrel Loading Dose | Prasugrel Maintenance Dose | Ticagrelor Maintenance Dose
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/41 | 1/35
Other Adverse Events (participants affected / at risk) | 8/34 | 10/41 | 12/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel Loading Dose (N=34) | Prasugrel Maintenance Dose (N=41) | Ticagrelor Maintenance Dose (N=35)
congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
depression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel Loading Dose (N=34) | Prasugrel Maintenance Dose (N=41) | Ticagrelor Maintenance Dose (N=35)
eccymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 4 (4)
headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
allergic oedema (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Consultants may not publish in any way without the prior written consent of Daiichi Sankyo Inc., which consent may be witheld by DSI in its sole discretion, any material or manuscript relating to Consultant's work hereunder and/or any information or materials that Consultant received in connection with or pursuant to this Agreement or Consultant's relationship established with DSI.